CLINICAL TRIAL: NCT06763445
Title: Exploring the Relationship Between Caring Experience, Perceived Behavioral Control, and Caring Intention Among University Students
Brief Title: Exploring the Relationship Between Caring Experience, Perceived Behavioral Control, and Caring Intention Among Students
Status: Recruiting | Type: Observational
Sponsor: Chiu Shu-Ching (Other)
Responsible Party: Sponsor-Investigator, Chiu Shu-Ching, Assistant Professor, Central Taiwan University of Science and Technology
Organization: Central Taiwan University of Science and Technology (Other)
Other Study IDs: CTU112JAH001
Record Dates: First submitted 2024-12-31; First posted 2025-01-08 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Caring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research project conducts a relevant investigation into the past background and learning experiences of university students during the process of caring. Additionally, it aims to understand the correlations between different scales.

ELIGIBILITY:
Inclusion Criteria:

* University students aged 18 and above.

Exclusion Criteria:

* University students who refuse or are unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: students
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
Caring Intention | Baseline. Will be collected only once.
  Score:1-80. A higher score means a better outcome.

SECONDARY OUTCOMES:
caring assessment scale | Baseline. Will be collected only once
  Score:1-100. A higher score means a better outcome.
Perceived Behavioral Control for caring | Baseline. Will be collected only once.
  Score:1-135. A higher score means a better outcome.
Caring Experience | Baseline. Will be collected only once.
  Score:1-250. A higher score means a better outcome.
caring ability inventory | Baseline. Will be collected only once.
  Score:1-259. A higher score means a better outcome.
Selfishness questionnaire | Baseline. Will be collected only once.
  Score:0-48. A lower score means a better outcome.
Scale for Measuring Changes in Ideas About Caring | Baseline. Will be collected only once.
  Score:1-135. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Taiwan University of Science and Technology, Taichung, Taiwan